CLINICAL TRIAL: NCT03054155
Title: Treatment of Hidradenitis Suppurativa With Eth 755nm Alexandrite Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Steven D Daveluy, Medical Doctor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 120116M1F
Record Dates: First submitted 2017-02-09; First posted 2017-02-15 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Hidradenitis Suppurativa
Keywords: hidradenitis suppurativa; hidradenitis; laser
MeSH Terms: conditions — Hidradenitis Suppurativa; Hidradenitis | interventions — Lasers, Solid-State

STUDY DESIGN:
Intervention Model Description: For each patient, one side of the body will serve as the treatment side and the other side as the control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment Arm (Experimental): For each patient, one side of the body will be treated with the Alexandrite laser (the treatment arm) and the other will not be treated to serve as control (the control arm). For example, if a patient has the disease in both axillae, one will treatment and the other control
  Interventions: Device: Alexandrite Laser
- Control Arm (No Intervention): For each patient, one side of the body will be treated with the Alexandrite laser (the treatment arm) and the other will not be treated to serve as control (the control arm). For example, if a patient has the disease in both axillae, one will treatment and the other control

INTERVENTIONS:
Device: Alexandrite Laser — Alexandrite 755nm hair removal laser
  Arms: Treatment Arm

SUMMARY:
Patients with bilateral hidradenitis in the axilla, groin and/or inframammary will be treated on one side with the Alexandrite hair removal laser. The other side will serve as the control.

DETAILED DESCRIPTION:
Patients with bilateral disease will be chosen to participate in the study. Patients will be advised to discontinue any prior systemic HS treatments two weeks before their first laser session as a wash out period. One side of the patient will be chosen as the treatment side, the other as an intrinsic control. Each participant will have a total of 4 treatments with the laser, one treatment per month over the duration of 4 months. Patients will then participate in a follow-up clinic visit two months after completion of their last treatment. In between laser sessions, participants will be allowed to use benzoyl peroxide 10% wash as a skin cleanser and clindamycin 1% solution or lotion as a topical therapy, both twice daily to the treatment and control areas. At each visit, photographs will be taken of the lesions to monitor progression and to serve as a comparison to the control side. The treatment side will be treated with the laser and adjusted according to skin type as follows:

Skin type I-II (Fair Caucasian): Fluence: 30J/cm2 Skin type III (Darker Caucasian, light Asian): Fluence: 25 J/cm2 Skin type IV (Mediterranean, Asian, Latin): Fluence: 18 J/cm2 Skin type V (Light skinned black, Darker mediterranean): Fluence: 16J/cm2 Skin type VI (Dark skinned black): Fluence 14 J/cm2

A spot size of 12 mm and a cryogen spray delay of 50/50 will be used for all treated patients. The treatment area will not exceed 15cm x 15cm. If the patient cannot tolerate treatment with the Alexandrite laser, the patient will be terminated from the study. Following each treatment session, the patient will be given an ice pack to reduce any discomfort the patient may experience as a result of treatment with the laser. Clinical evaluation and photographs will determine improvement.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Patients with Hidradenitis Suppurativa with bilateral and symmetric disease with one or more anatomic sites of involvement.

Exclusion Criteria:

* Pregnant patients or patients planning to get pregnant during the time of the study
* Patients on systemic treatment for Hidradenitis Suppurativa
* Patients with photosensitivity disorders
* Patients unable to tolerate the laser treatments
* Intake of a photosensitive medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
HS-LASI | Monthly for 4 months, then once 2 months later(6 months total)
  Change in Hidradenitis Suppurativa Lesion, Area, and Severity Index Score from baseline

SECONDARY OUTCOMES:
HiSCR | Monthly for 4 months, then once 2 months later(6 months total)
  Change in Hidradenitis Suppurativa Clinical Response Scale from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne State University Physician Group Dermatology, Dearborn, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tierney E, Mahmoud BH, Hexsel C, Ozog D, Hamzavi I. Randomized control trial for the treatment of hidradenitis suppurativa with a neodymium-doped yttrium aluminium garnet laser. Dermatol Surg. 2009 Aug;35(8):1188-98. doi: 10.1111/j.1524-4725.2009.01214.x. Epub 2009 May 12. PMID 19438670
- [Background] Mahmoud BH, Tierney E, Hexsel CL, Pui J, Ozog DM, Hamzavi IH. Prospective controlled clinical and histopathologic study of hidradenitis suppurativa treated with the long-pulsed neodymium:yttrium-aluminium-garnet laser. J Am Acad Dermatol. 2010 Apr;62(4):637-45. doi: 10.1016/j.jaad.2009.07.048. PMID 20227579
- [Background] Kimball AB, Sobell JM, Zouboulis CC, Gu Y, Williams DA, Sundaram M, Teixeira HD, Jemec GB. HiSCR (Hidradenitis Suppurativa Clinical Response): a novel clinical endpoint to evaluate therapeutic outcomes in patients with hidradenitis suppurativa from the placebo-controlled portion of a phase 2 adalimumab study. J Eur Acad Dermatol Venereol. 2016 Jun;30(6):989-94. doi: 10.1111/jdv.13216. Epub 2015 Jul 22. PMID 26201313